CLINICAL TRIAL: NCT05664295
Title: Comparison of Plasma Orexin-A Levels and Awakening Time From Anesthesia in Patients With and Without Insomnia Who Had Laparoscopic Cholecystectomy Under General Anesthesia
Brief Title: Orexin-A Levels in Insomnia Patients
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Melike Korkmaz Toker, Associate Professor of Anesthesiology and Reanimation, Muğla Sıtkı Koçman University
Other Study IDs: 14/III
Record Dates: First submitted 2022-11-21; First posted 2022-12-23 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Insomnia; Anesthesia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- insomnia patients: Jenkins Sleep Disorders scale skor >1 and Epworth Sleepiness scale skor >9
  Interventions: Diagnostic Test: Jenkins Sleep Disorders scale and Epworth Sleepiness scale
- noninsomniacs: Jenkins Sleep Disorders scale skor <2 and Epworth Sleepiness scale skor <10
  Interventions: Diagnostic Test: Jenkins Sleep Disorders scale and Epworth Sleepiness scale

INTERVENTIONS:
Diagnostic Test: Jenkins Sleep Disorders scale and Epworth Sleepiness scale — Jenkins Sleep Disorders scale and Epworth Sleepiness scale

SUMMARY:
In the pathophysiology of insomnia, the increase of the orexin-A (OXA) peptide released from orexin neurons in the lateral hypothalamus plays an important role. Orexins takes part at the emergence of anesthesia. In the literature, investigators could not attain any studies about the arousal of insomnia patients from anesthesia. In this study, the effect of this peptide on the emergence process from anesthesia was investigated by comparing plasma OXA levels before and after anesthesia in insomnia patients.

DETAILED DESCRIPTION:
ASA (American Society of Anesthesiologists) I-II patients aged 18-65 years who underwent elective laparoscopic cholecystectomy were included in the study. Patients were evaluated with the Jenkins Sleep Disorders scale and Epworth Sleepiness scale during preoperative examination and were divided into insomnia and control groups. Blood samples were obtained for OXA and glucose levels at anesthesia induction, 5 minutes after extubation and 30 minutes after extubation. The times from stopping anesthesia to eyes opening and extubation and end-tidal sevoflurane concentrations at these time points were recorded.

ELIGIBILITY:
Inclusion Criteria:

* male patients undergo elective laparoscopic cholecystectomy under general anesthesia
* Between 18-65 age
* ASA I-II

Exclusion Criteria:

* ASA≥III
* Patients with obstructive sleep apnea syndrome
* Bleeding over 500 ml
* Allergic to anesthetic agents
* Patients with a BMI > 30 kg/m2

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Study Population: Male patients undergo elective laparoscopic cholecystectomy under general anesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Orexin-A Levels | at anesthesia induction, 5 minutes after extubation and 30 minutes after extubation
  plasma OXA levels anesthesia induction and after anesthesia in insomnia patients
Orexin-A Levels | at anesthesia induction, 5 minutes after extubation and 30 minutes after extubation
  plasma OXA levels anesthesia induction and after anesthesia in control group

SECONDARY OUTCOMES:
recovery time from general anesthesia | time of eyes opening and time of extubation
  The relationship between plasma OXA levels and recovery times from anesthesia in insomnia patients

CONTACTS AND LOCATIONS:
Overall Officials: melike Korkmaz Toker, Principal Investigator — Mugla Sıtkı Kocman University Department of Anesthesiology and reanimation
Locations (1):
- Mugla Sitki Kocman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bollu PC, Kaur H. Sleep Medicine: Insomnia and Sleep. Mo Med. 2019 Jan-Feb;116(1):68-75. PMID 30862990
- [Background] Hirota K. [Orexinergic neurons and noradrenergic awakening system in general anesthesia]. Masui. 2007 Jan;56(1):9-18. Japanese. PMID 17243641
- [Background] Erden V, Abitagaoglu S, Guler C, Dogan Z, Kirgezen S, Abut Y. Insomnia may increase anesthetic requirement. J Clin Anesth. 2016 Nov;34:367-72. doi: 10.1016/j.jclinane.2016.05.020. Epub 2016 Jun 4. No abstract available. PMID 27687412